CLINICAL TRIAL: NCT00611195
Title: Impact of Remifentanil Administration on Laryngeal Reflex Responses in Pediatric Patients With Upper Respiratory Anesthetized With Propofol
Brief Title: Remifentanil and Laryngeal Reflex Responses in Pediatric Patients With URI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Erb (Other)
Responsible Party: Sponsor-Investigator, Thomas Erb, Prof.Dr. Thomas Erb, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UNIBAS:UKBB_ANE_LR5; SNF3200B0-109322 (Other: SNF 3200B0-109322)
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Upper Respiratory Infections
Keywords: Anesthesia; Children; Larynx
MeSH Terms: conditions — Respiratory Tract Infections; Laryngeal Diseases | interventions — Propofol; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Larynx assessment under stimulation
  Interventions: Drug: propofol, remifentanil

INTERVENTIONS:
Drug: propofol, remifentanil — propofol 3micrgr/ml (TCI plasma concentration Kataria model) versus propofol 3micrgr/ml and remifentanil 0.05microgr/kg/min
  Other Names: Recofol; Disoprivan; Ultiva

SUMMARY:
To describe respiratory and laryngeal responses to laryngeal stimulation during propofol anesthesia in children with upper airway infections. To determine whether the co-administration of remifentanil blunts these reflex responses. To test whether the co-administration of remifentanil results in a significant reduction of apnea with laryngospasm in these patients.

Hypotheses:

I: In children with a URI undergoing anesthesia with propofol, the incidence of apnea and laryngospasm after controlled stimulation is expected to occur 2.5 times more frequently than in children without URI (20 vs. 8%).

II: The incidence of apnea and laryngospasm is diminished after administration of remifentanil.

DETAILED DESCRIPTION:
Patients undergoing anesthesia in the presence of an upper respiratory infection (URI) are very common in pediatric anesthesia practice. Although, clinical data confirm that children with URIs are at increased risk of perioperative complications, it has become standard practice not to postpone anesthesia in the presence of URI. While complications (such as cough, hypoxemia) can be anticipated, recognized, and treated, laryngospasm remains the most severe and dramatic complication. In clinical practice, patients who develop laryngospasm are greater than 2.5 times more likely to have an active upper respiratory infection; therefore, knowledge that allows for rational selections of anesthetic agents under this condition is highly warranted. Based on our results obtained in healthy children, the use of propofol appears to be most promising under these circumstances. For this reason, the laryngeal and respiratory reflex responses should be assessed in patients with URI anaesthetized with propofol.

Commonly held believes suggest, that the administration of opioids blunts airway reflexes, including laryngospasm. However, in a previous study of our group in children anesthetized with sevoflurane the administration of fentanyl effectively blunted all airway reflexes but laryngospasm. These results are in contrast to those obtained in adults anesthetized with propofol where fentanyl also effectively blunted laryngospasm.

In children the combined use of propofol and remifentanil has become more frequent, particularly because of its synergistic pharmacodynamic effect. Besides its use during surgical procedures, this regime is also being increasingly advocated for diagnostic procedures such as bronchoscopy and esophago-gastroduodenoscopy. These interventions include instrumentation of the airway in children that are at an increased risk of harmful effects of laryngeal reflex responses.

Despite their obvious clinical significance, reflexes that involve the function of the upper airway are only minimally understood and information on such reflexes is scarce in anesthetized humans. Nonetheless, a model was developed by analyzing respiratory variables and endoscopic images after stimulating the laryngeal mucosa with a small amount of distilled water. This model was successfully adapted to the pediatric setting by our group assessing the impact of propofol, sevoflurane, fentanyl and lidocaine administration on laryngeal reflex responses in preschool children.

ELIGIBILITY:
Inclusion Criteria:

* ASA I + II
* elective intervention under general anesthesia
* acute upper respiratory tract infection

Exclusion Criteria:

* chronic respiratory tract infection
* fever >38,3° celsius
* productive cough
* neuromuscular disease
* malignant hyperthermia
* cardiac disease

Ages: 25 Months to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2008-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Occurence of laryngospasm (defined as complete closure of the vocal or false cords with apnea lasting >10sec) after laryngeal stimulation | 5min

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O Erb, MD, Principal Investigator — Universitiy children's hospital Basel
Locations (1):
- University children's hospital, Basel, Switzerland

REFERENCES:
- [Background] Oberer C, von Ungern-Sternberg BS, Frei FJ, Erb TO. Respiratory reflex responses of the larynx differ between sevoflurane and propofol in pediatric patients. Anesthesiology. 2005 Dec;103(6):1142-8. doi: 10.1097/00000542-200512000-00007. PMID 16306725